CLINICAL TRIAL: NCT05907720
Title: Evaluation of Prototype Solutions in Improving Uptake and Adherence to Institutional Delivery, ANC, and IFA Supplementation Services Among Pregnant Women in Selected Woredas of Ethiopia
Brief Title: Evaluation of Prototype Solutions for Optimizing Maternal Health Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00024473
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Maternal Behavior
Keywords: Birth Setting; Prenatal Care; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention arm will receive a package of behavioral interventions in addition to usual care in health facilities.
  Interventions: Behavioral: Human-centered design prototype solutions for vulnerable pregnant women
- Control Arm (No Intervention): The control arm will not receive any intervention other than usual care.

INTERVENTIONS:
Behavioral: Human-centered design prototype solutions for vulnerable pregnant women — The intervention package will include various social and behavior change programs derived from a human-centered design approach. The intervention will be tailored to vulnerable pregnant women's needs and contexts. It may include but is not limited to health communication campaigns, including radio and print media.
  Arms: Intervention Arm

SUMMARY:
This study is a three-year implementation research project that aims to develop and test the effectiveness and acceptability of interventions to promote three outcomes: institutional delivery, antenatal care, and iron-folic acid supplementation among pregnant women in Ethiopia. The project applies a Human-Centered-Design (HCD) to develop prototype solutions that optimize the uptake and adherence to maternal and child health services by pregnant women. The evaluation of high-fidelity prototype solutions that come out from a sprint workshop (rapid HCD) and an extended HCD process will take place across two phases.

DETAILED DESCRIPTION:
With funding and support from the Bill and Melinda Gate Foundation (BMGF), a three-year implementation research project will be conducted to develop and test the effectiveness and acceptability of interventions to promote three outcomes: institutional delivery, antenatal care (ANC) and iron folic acid (IFA) supplementation among pregnant women. The project applies a Human-Centered-Design (HCD) to develop prototype solutions that optimize the uptake of and adherence to maternal and child health services by pregnant women. Initial and high-fidelity prototype solutions that come out from a sprint workshop (rapid HCD) and an extended HCD process will be implemented in two phases.

Phase 1: The investigators will conduct a design sprint workshop and develop prototype solutions focusing on ANC and institutional delivery and the high-fidelity prototypes will be implemented for four months. The prototype solutions may include but are not limited to social and behavior change communication campaigns, including print media, mass media, social media, and community-based educational events. Specific content and format of the prototypes will be determined based on participant needs and preferences identified from the workshop. Baseline and midline assessments will be conducted to evaluate the effectiveness of the prototypes.

Phase 2: The investigators will conduct extended HCD to refine prototype solutions for design challenges around ANC and institutional delivery that are not addressed by the design sprint. The prototype solutions may include but are not limited to social and behavior change communication campaigns, including print media, mass media, social media, and community-based educational events. Specific content and format of the prototypes will be determined based on participant needs and preferences identified from the workshops in Phases 1 and 2. High-fidelity prototypes designed in the two phases will be implemented in the two intervention Woredas (geographical areas in Ethiopia roughly equivalent to counties in the US) for another four months. A post-intervention cross-sectional assessment will be conducted to evaluate the effectiveness of the prototypes.

Hence, the following four research activities will occur throughout the study: (1) baseline in Year 1 and (2) midline in Year 1, possibly bleeding into Year 2. These two waves will involve the same pregnant women recruited at baseline. (3) end-line in Year 3; this last assessment will recruit newly pregnant women to compare with the recruited panel at baseline. All rounds of evaluations (three data waves in total) have the objective of assessing the effectiveness of the intervention in improving (a) institutional delivery and (b) uptake of ANC services. In addition, qualitative interviews will assess psychosocial and intermediate outcomes among pregnant women as well as implementation research outcomes of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant 5+ months
* 15 to 49 years
* moderate to high vulnerability

Exclusion Criteria:

* Pregnant less than 5 months
* non-reproductive age
* low vulnerability

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1024 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in institutional delivery rates assessed by the survey instrument | Baseline and 4 months
  Institutional delivery will be measured using a question that asks about a place of child birth in most recent pregnancy
Change in the number of antenatal care visits assessed by the survey instrument | Baseline and 4 months
  The outcome will be measured using a question that asks about the number of antenatal care visits women had during current pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Rimal, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Communication Programs, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a publication will be shared after deidentification. The data will be shared with researchers whose proposed use of the data has been approved by an independent review committee for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.